CLINICAL TRIAL: NCT00005392
Title: Epidemiology of Venous Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4298; R01HL053487 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2005-07

CONDITIONS: Cardiovascular Diseases; Peripheral Vascular Diseases; Telangiectasis
MeSH Terms: conditions — Cardiovascular Diseases; Peripheral Vascular Diseases; Telangiectasis

SUMMARY:
To conduct several studies on the epidemiology of venous disease.

DETAILED DESCRIPTION:
BACKGROUND:

Venous disease is commonplace, more prevalent in women, increases with age, and is a major cause of morbidity. Between 6 and 30 percent of all medical expenditures for cardiovascular disease are for venous disease. Despite these facts, the basic epidemiology of venous disease has received limited attention. Even the definition of peripheral venous disease varies widely, often confusing symptoms and signs with demonstrable pathophysiologic abnormalities.

This study provided estimates of the extent of peripheral venous disease, contributed to more efficient diagnosis, allowed insight on how to prevent or ameliorate this condition through risk factor modification, and provided quantitative estimates of the daily burden this disease imposes on patients.

DESIGN NARRATIVE:

The overall, and age, sex, and ethnic-specific, prevalence of peripheral venous disease was determined in a stratified multiethnic random sample of 2,408 men and women aged 29 to 91 years. Three specific categories of venous disease were defined including: telangiectasias and flat reticular veins; superficial venous disease without deep valvular incompetence or obstruction; deep venous disease, with valvular incompetence or obstruction. Varicose veins were typically but not invariably present in the latter two categories. These three categories were diagnosed by an ordered non-invasive evaluation, including visual inspection, with photographic documentation of abnormal findings, and duplex color sonography to diagnose valvular incompetence and venous obstruction.

An evaluation was made of the sensitivity, specificity, and predictive value of each of the traditional signs and symptoms of venous disease for each of the three categories of venous disease. Signs and symptoms evaluated included aching, itching, swelling and edema, heaviness, cramps, nocturnal restless legs, pigmentation, induration, ulcers, and the Trendelenburg test. Risk factors were evaluated for each of the above three categories-of venous disease. Risk factors assessed included age; sex; ethnicity; socioeconomic status; height; weight; obesity; exercise; blood pressure; standing versus sitting in daily activities; family history of venous disease; cigarette smoking; alcohol consumption; diet; constipation; constrictive clothing; aspirin use; use of selected other medications; history of hernia, flat feet, or other conditions associated with connective tissue laxity; parity; use of estrogens or progestins; age at menarche; age at menopause; and concomitant arterial disease. Finally, an evaluation was made of the degree of morbidity and interference with daily activities resulting from venous disease, using the Quality of Well Being (QWB) scale developed at University of California at San Diego.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 29 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1995-09; Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Criqui — University of California, San Diego

REFERENCES:
- [Background] Fronek A, Criqui MH, Denenberg J, Langer RD. Common femoral vein dimensions and hemodynamics including Valsalva response as a function of sex, age, and ethnicity in a population study. J Vasc Surg. 2001 May;33(5):1050-6. doi: 10.1067/mva.2001.113496. PMID 11331848
- [Background] Langer RD, Ho E, Denenberg JO, Fronek A, Allison M, Criqui MH. Relationships between symptoms and venous disease: the San Diego population study. Arch Intern Med. 2005 Jun 27;165(12):1420-4. doi: 10.1001/archinte.165.12.1420. PMID 15983292
- [Background] Criqui MH, Jamosmos M, Fronek A, Denenberg JO, Langer RD, Bergan J, Golomb BA. Chronic venous disease in an ethnically diverse population: the San Diego Population Study. Am J Epidemiol. 2003 Sep 1;158(5):448-56. doi: 10.1093/aje/kwg166. PMID 12936900